CLINICAL TRIAL: NCT07370610
Title: Electrical Impedance Tomography-Based Dynamic Ventilation-Perfusion Functional Phenotype Trajectory in Acute Respiratory Distress Syndrome: A Prospective Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20250516
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: ARDS; Mechanically Ventilated Patients
Keywords: eit; lung perfusion patterns; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EIT Monitoring group: * 16-electrode belt positioned around the thorax
  * Daily perfusion assessment (10 min recording) at baseline and after major clinical interventions (e.g., PEEP change, position change)
  * Pulmonary perfusion analysis will primarily be based on the pulse-synchronous impedance signal derived from EIT during brief respiratory pauses, estimating regional perfusion from cardiac-related impedance changes. When signal quality is insufficient, or in cases of significant arrhythmia or other conditions affecting pulse signal detection, the saline indicator method will be applied for validation or calibration.
  * This involves rapid intravenous bolus injection of 10-20 mL room-temperature saline, using the induced transient conductivity change as a perfusion marker:Ventilation-Perfusion Functional Phenotype will be derived by combining EIT-based tidal and pulsatile impedance changes, calculating the regional V/Q ratio.
  Interventions: Device: EIT Monitoring

INTERVENTIONS:
Device: EIT Monitoring — * 16-electrode belt positioned around the thorax
  * Daily perfusion assessment (10 min recording) at baseline and after major clinical interventions (e.g., PEEP change, position change)
  * Pulmonary perfusion analysis will primarily be based on the pulse-synchronous impedance signal derived from EIT during brief respiratory pauses, estimating regional perfusion from cardiac-related impedance changes. When signal quality is insufficient, or in cases of significant arrhythmia or other conditions affecting pulse signal detection, the saline indicator method will be applied for validation or calibration.
  * This involves rapid intravenous bolus injection of 10-20 mL room-temperature saline, using the induced transient conductivity change as a perfusion marker:Ventilation-Perfusion Functional Phenotype will be derived by combining EIT-based tidal and pulsatile impedance changes, calculating the regional V/Q ratio.

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is characterized by severe hypoxemia and extensive lung injury. Recent studies indicate that lung functional phenotypes - particularly the distribution and evolution of lung perfusion - may be closely related to patient outcomes. Electrical impedance tomography (EIT) offers non-invasive, bedside, real-time monitoring of lung perfusion patterns and enables classification into distinct phenotypes and trajectory types over the course of illness. To date, limited data exist on perfusion phenotype trajectories in ARDS patients and their relationship with clinical outcomes. This study seeks to characterize dynamic lung dynamic ventilation-perfusion functional Phenotype using EIT and explore their prognostic significance. Objectives

Primary Objective:

To identify lung perfusion phenotype trajectories in ARDS patients using EIT and assess their association with 28-day mortality.

Secondary Objectives:

* To determine the relationship between different trajectory types and improvements in oxygenation and respiratory mechanics.
* To investigate how ventilator settings (PEEP, driving pressure) interact with perfusion changes.
* To support individualized mechanical ventilation strategies based on Ventilation-Perfusion Functional Phenotype monitoring

DETAILED DESCRIPTION:
Design: Prospective, multicenter, observational cohort study

* Setting: ≥2 tertiary ICUs equipped with EIT capability
* Population: Adult patients with moderate-to-severe ARDS (Berlin definition, PaO₂/FiO₂ ≤ 200 mmHg) receiving mechanical ventilation
* Intervention: Daily lung perfusion assessment using a 16-electrode EIT belt. Regional ventilation-perfusion (V/Q) ratios are calculated by combining tidal and pulsatile impedance changes. Phenotypes are classified as Matched V/Q, High V/Q (dead space), Low V/Q (shunt), or Globally Impaired V/Q. Trajectories are categorized as Stable, Improving, Deteriorating, or Fluctuating.
* Endpoints:
* Primary: Association between phenotype trajectory type and 28-day mortality
* Secondary: Time to oxygenation improvement, duration of mechanical ventilation, ICU length of stay, interaction between trajectory and ventilator settings

ELIGIBILITY:
Inclusion Criteria:

* ge ≥ 18 years
* Moderate-to-severe ARDS (Berlin definition, PaO₂/FiO₂ ≤ 200 mmHg)
* Mechanically ventilated and eligible for EIT monitoring
* Informed consent obtained from patient or legal surrogate

Exclusion Criteria:

* Pregnancy
* Presence of implanted metallic devices interfering with EIT (e.g., pacemaker)
* Severe chest wall deformity or skin condition preventing electrode placement
* Expected survival < 24 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS Mechanically Ventilated Patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | From enrollment to 28 days

SECONDARY OUTCOMES:
Time to oxygenation improvement (PaO₂/FiO₂ > 200 mmHg) | From enrollment until the event occurs, assessed up to 14 days
Duration of mechanical ventilation | From intubation until successful extubation, assessed up to 28 days or until ICU discharge/death
ICU length of stay | From ICU admission until discharge from ICU, assessed up to 60 days
Interaction between phenotype trajectory and ventilator settings (PEEP, driving pressure) | Daily during EIT monitoring period, up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Qu, Study Chair — Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided